CLINICAL TRIAL: NCT06169865
Title: Prevalence of Peripheral Vascular Diseases and Presentation in Patients With Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hossam Adly Mohamed (Other)
Responsible Party: Sponsor-Investigator, Hossam Adly Mohamed, resident at vascular surgery department, Sohag University
Organization: Sohag University (Other)
Other Study IDs: soh-Med-23-10-03MS
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Vascular Diseases and Presentation in Patient With Autoimmune Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cross sectional study — cross sectional study to explore magnitude of peripheral vascular diseases and presentations in patients with autoimmune diseases in sohag society.

SUMMARY:
Rheumatic autoimmune diseases include conditions such as systemic lupus rheumatoid arthritis systemic sclerosis in which connective tissues are frequently targeted.

Autoimmune diseases as a group are among the leading causes of death and morbidity in the industrial world and pose an immense socioeconomic burden despite the considerable accumulative burden of these diseases only a small number of multinational registries for a few selected autoimmune diseases have been devised.

Numerous autoimmune inflammatory diseases have been associated with various forms of vasculopathy and increase vascular disease risk such as accelerated atherogenesis and thromboembolic events as digital and acral gangrene secondary Raynaud syndrome arterial aneurysm and different cutaneous ulcer.

The etiopathogenesis os increased risk of peripheral vascular diseases and presentation in autoimmune diseases is not entirely clear but multiple contibutors have been explored especially in the context of systemic inflammation and disordered thrombogenesis.

ELIGIBILITY:
Inclusion Criteria:

* all ages
* Both sexes
* Recent or past history of vascular diseases or presentation in any proven autoimmune diseases according to the guidlines.

Exclusion Criteria:

* patients refuse the study
* patients do not have established diagnosis of vascular diseases .
* patients not completely approved to have autoimmune diseases.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * All ages
  * Both sexes
  * Recent or past history of vascular diseases or presentation in any proven autoimmune diseases according to the guidlines.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
prevalence of peripheral vascular diseases and presentations in patients with autoimmune diseases . | 6 months
  old and new vascular diseases and presentations in patients with autoimmune diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Cooper GS, Bynum ML, Somers EC. Recent insights in the epidemiology of autoimmune diseases: improved prevalence estimates and understanding of clustering of diseases. J Autoimmun. 2009 Nov-Dec;33(3-4):197-207. doi: 10.1016/j.jaut.2009.09.008. Epub 2009 Oct 9. PMID 19819109
- [Background] Zoller B, Li X, Sundquist J, Sundquist K. Autoimmune diseases and venous thromboembolism: a review of the literature. Am J Cardiovasc Dis. 2012;2(3):171-83. Epub 2012 Jul 25. PMID 22937487
- [Background] Bashal F. Thrombosis in Rheumatological Diseases. 2021 Jan 6. In: Almoallim H, Cheikh M, editors. Skills in Rheumatology [Internet]. Singapore: Springer; 2021. Chapter 12. Available from http://www.ncbi.nlm.nih.gov/books/NBK585742/ PMID 36315801
- [Background] Pyrpasopoulou A, Chatzimichailidou S, Aslanidis S. Vascular disease in systemic lupus erythematosus. Autoimmune Dis. 2012;2012:876456. doi: 10.1155/2012/876456. Epub 2012 Aug 22. PMID 22957213